CLINICAL TRIAL: NCT03626779
Title: Prf Controlled,Randamized Cinical Trial of EFFECTS OF THE PLATELET-RICH FIBRIN (PRF) ON BONE DENSITY IN IMMEDIATE IMPLANT PLACEMENT AND LOADING IN ESTHETIC ZONE
Brief Title: Bone Density in Immediate Implant Placment and Loading(BDIIPL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed adel shaaban (Other)
Responsible Party: Sponsor-Investigator, Ahmed adel shaaban, CairoU, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo U
Record Dates: First submitted 2018-07-30; First posted 2018-08-13 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Bone Density Increased
MeSH Terms: conditions — Osteosclerosis | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate placment and loading with prf (Other): Immediat placment and loading with prf
  Interventions: Other: Prf
- immediate implant placment and loading (No Intervention): Immediate implant placment and loading without prf

INTERVENTIONS:
Other: Prf — Take 10cc blood from patient and gain prf blug
  Arms: immediate placment and loading with prf

SUMMARY:
Atrumatic extraction ,immediate implant placment , prf as plug,immediate loading , mesure bone density 0-3-6-9 month

DETAILED DESCRIPTION:
Atrumatic extraction unrestorable tooth in esthetic zone and immediate implant placment and withdrow 10cc blood sample to gain prf plug as membrane and immediate provisional for one week and final restoration after 1 week , and mesure bone density from 0-3-6-9 month

ELIGIBILITY:
Inclusion criteria:

* unrestorable anterior tooth.
* Good oral hygine
* Adequate bone hieght apical to the alveolus of failing tooth to ensure primary stability .

Exclusion Criteria:

* systematic disease which affect osteointgration.
* Bad oral hygiene
* Broxism, clenching, deep bite, edge to edge and abnormal habits.
* Non-treated peeiodontal diseases.
* Pregnancy and smokers. Severe infection. Loss of labial crest after extraction of failing tooth.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Bone density enhancement with prf in immediate implant placment and loding | 9 month
  Cbct